CLINICAL TRIAL: NCT02183636
Title: Relative Bioavailability of Two Fixed Dose Combination Tablets of Linagliptin 5 mg/Pioglitazone 45 mg Compared With Single Linagliptin 5 mg and Pioglitazone 45 mg Tablets Administered Together to Healthy Male and Female Subjects (Open, Randomised, Single Dose, Three-period Crossover Phase I Trial)
Brief Title: Relative Bioavailability of Two Fixed Dose Combination Tablets of Linagliptin/Pioglitazone Compared With Single Linagliptin and Pioglitazone Tablets Administered Together to Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1264.1
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Pioglitazone

ARMS (3):
- Treatment 1 (T1) (Experimental): Linagliptin/pioglitazone, FDC formulation C5
  Interventions: Drug: Linagliptin/pioglitazone, FDC formulation C5
- Treatment 2 (T2) (Experimental): Linagliptin/pioglitazone, FDC formulation C8
  Interventions: Drug: Linagliptin/pioglitazone, FDC formulation C8
- Reference (R) (Active Comparator): Linagliptin tablet and pioglitazone tablet (Actos®)
  Interventions: Drug: Linagliptin tablet; Drug: pioglitazone tablet (Actos®)

INTERVENTIONS:
Drug: Linagliptin/pioglitazone, FDC formulation C5 — film coated tablet (5 mg/45 mg)
  Arms: Treatment 1 (T1)
Drug: Linagliptin/pioglitazone, FDC formulation C8 — film coated tablet (5 mg/45 mg)
  Arms: Treatment 2 (T2)
Drug: Linagliptin tablet — 5 mg
  Arms: Reference (R)
Drug: pioglitazone tablet (Actos®) — 45 mg
  Arms: Reference (R)

SUMMARY:
Determination of the relative bioavailability of 2 different formulations of a 5 mg linagliptin (BI 1356)/45 mg pioglitazone fixed dose combination (FDC) tablet, formulation C5 and formulation C8, compared with the mono-components linagliptin and pioglitazone administered together

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects according to the following criteria: based upon a complete medical history, including physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age ≥18 and ≤55 years
* Body mass index (BMI) ≥18.5 and ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy), psychiatric disorders, or neurological disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 h) within at least 1 month or less than 10 halflives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day for males and 20 g/day for females)
* Drug abuse
* Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site

For female subjects:

* Pregnancy or a positive pregnancy test, planning to become pregnant during the study, or within 1 month of study completion or lactation period
* No adequate contraception during the study and until 1 month after study completion, i.e. implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence (for at least 1 month before enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females who did not have a vasectomised partner, were not sexually abstinent, or were not surgically sterile were asked to additionally use barrier contraception methods (i.e. condom, diaphragm with spermicide)

For male subjects:

* Male subjects who did not agree to minimise the risk of female partners becoming pregnant from the first dosing day until the completion of the post study medical examination. Acceptable methods of contraception included barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive for at least 2 months)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUC0-72 (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 to 72 h) | 1 hour prior drug administration and up to 120 h after drug administration
Cmax (maximum measured concentration of linagliptin in plasma) | 1 hour prior drug administration and up to 120 h after drug administration
AUC0-infinity (area under the concentration-time curve of pioglitazone in plasma over the time interval from 0 extrapolated to infinity) | 1 hour prior drug administration and up to 72 h after drug administration
Cmax (maximum measured concentration of pioglitazone in plasma) | 1 hour prior drug administration and up to 72 h after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | 1 hour prior drug administration and up to 120 h after drug administration
AUC0-infinity (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 extrapolated to infinity) | 1 hour prior drug administration and up to 120 h after drug administration
AUC0-72 (area under the concentration-time curve of pioglitazone in plasma over the time interval from 0 to 72 h) | 1 hour prior drug administration and up to 72 after drug administration
Changes from baseline in vital signs (blood pressure (BP) and pulse rate (PR)) | 21 to 1 day prior start of treatment, at study visits 2 to 4 (prior to treatment administration and 24 h following treatment administration), and 7 days after last treatment administration
Occurrence of adverse events (AEs) | until 7 days after last treatment administration
Assessment of tolerability by the investigator | on day 6 of each treatment and 7 days after last treatment administration